CLINICAL TRIAL: NCT04362228
Title: The Effects of Whole-body Exercise to Improve Swallowing Function in Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Joseph Brant Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB project #10638
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Old Age; Dementia; Swallowing Disorder; Cough; Parkinson Disease; Neuro-Degenerative Disease
Keywords: dementia; swallowing; physical exercise; parkinson disease
MeSH Terms: conditions — Alzheimer Disease; Deglutition Disorders; Cough; Parkinson Disease; Dementia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-body exercise (Experimental)
  Interventions: Behavioral: Whole-body exercise

INTERVENTIONS:
Behavioral: Whole-body exercise — 10-week one-on-one, virtual, whole-body exercise class, 3x/week, focused on increasing respiratory rate through moderate-intensity aerobic exercises.

SUMMARY:
Swallowing impairment (dysphagia) is extremely common in older adults living with dementia due to age-related changes in swallowing and other disease-specific impairments. Dysphagia is commonly managed by modifying diet textures rather than engaging in rehabilitative swallowing therapy. This means that countless people with dementia are left to eat pureed foods and drink thickened liquids, which are unpalatable and lead to malnutrition. As the disease progresses, many are transferred to nursing homes. In Canada, speech-language pathologists, who manage dysphagia, are consultants within nursing homes; therefore, swallowing therapy is non-existent. However, exercise therapy is more commonly available. Rodent models have demonstrated that physical exercise strengthens tongue and vocal-fold musculature, which are critical components of swallowing. Therefore, it is possible that whole-body physical exercise, which increases rate of respiration, will help to strengthen swallowing-related musculature in older adults with dementia. In this study, older adults (65+) with early-stage dementia will complete a 12-week physical exercise program to determine improvement of swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* > 59 years of age
* able to walk independently with or without an assistive device for a distance of at least 10 meters
* able to be active for 60 minutes with rest breaks
* abe to independently follow directions
* not involved in active rehabilitation
* a diagnosis of a progressive neurologic disease
* a maximum value for tongue strength <40 kPa

Exclusion Criteria:

* neurological conditions other than a progressive neurologic disease
* significant cardiovascular conditions
* severe aphasia
* pain, other medical conditions or behavioural issues that would limit safe participation in the exercise program
* individuals with known structural causes of dysphagia
* individuals with known allergies to latex
* individuals receiving swallowing rehab

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in respiratory function from baseline to end of intervention | baseline, week 4, week 14 and week 16
  Measure via peak cough flow using a peak flow meter
Change in swallowing function from baseline to end of intervention | baseline, week 4, week 14 and week 16
  Measure via isometric tongue strength using an Iowa Oral Performance Instrument

SECONDARY OUTCOMES:
Change in aerobic fitness from baseline to end of intervention | baseline, week 4, week 14 and week 16
  Measure via physical capacity using the 6-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kletzien H, Russell JA, Connor NP. The effects of treadmill running on aging laryngeal muscle structure. Laryngoscope. 2016 Mar;126(3):672-7. doi: 10.1002/lary.25520. Epub 2015 Aug 8. PMID 26256100
- [Background] Kletzien H, Russell JA, Leverson GE, Connor NP. Differential effects of targeted tongue exercise and treadmill running on aging tongue muscle structure and contractile properties. J Appl Physiol (1985). 2013 Feb 15;114(4):472-81. doi: 10.1152/japplphysiol.01370.2012. Epub 2012 Dec 20. PMID 23264540